CLINICAL TRIAL: NCT02683304
Title: S100B Protein Measures in the Care of Non-traumatic Headaches in the Emergency Department
Brief Title: S100B in the Care of Non-traumatic Headaches in the Emergency Department
Acronym: S100B-Céph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2015/RGG-01; 2016-A00013-48 (Other: ANSM)
Record Dates: First submitted 2016-01-19; First posted 2016-02-17 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2020-07

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study population (Experimental): The study population consists of consecutive headache patients (visual analogue scale > 3) presenting at the emergency department of the Nîmes University Hospital
  Interventions: Biological: Plasma S100B levels at inclusion; Device: Magnetic resonance imaging

INTERVENTIONS:
Biological: Plasma S100B levels at inclusion — Patients will have blood drawn to measure plasma S100B levels at inclusion.
Device: Magnetic resonance imaging — If not performed under emergency conditions, patients will have an MRI on days 2-4.

SUMMARY:
The main objective of this pilot study is to make a first assessment of the discriminating ability of a dosage of S100B protein for differential diagnosis between primary headaches and secondary headaches.

For this, the investigators will compare serum S100B protein between two groups of headache patients presenting at the emergency department: 1 group of primary headache patients and 1 group of secondary headache patients.

If the difference between the two groups proves potentially discriminating, the investigators will seek to determine the discriminating ability of the S100B protein by calculating the area under the ROC curve.

The reference diagnostic will be set at one month across the entire clinical picture and imaging by an expert committee composed of a neurologist, a radiologist and an emergency physician.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To seek an association between S100B protein levels and the onset of pain depending on whether it is more or less than 3 hours.

B. To assess the association between S100B protein levels and mortality at day 28.

C. To evaluate the association between S100B protein levels and hospital care: average length of stay in the emergency department, lumbar puncture, brain imaging, average length of hospital stay.

D. To evaluate the prognostic value of determination of S100B protein on the occurrence of a secondary headache at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has nontraumatic headache pain with a visual analog scale > 3

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication for magnetic resonance imaging
* Patients suffering from the following diseases: Alzheimer's disease, multiple sclerosis, Creutzfeldt-Jakob disease, melanoma, trisomy 21.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
S100B protein level (ng/ml) | Day 0
The presence/absence of a clinically significant anomaly on the MRI scan | Days 2-4
Final diagnostic as established by an expert committee | Month 1
  The diagnostic posed is either "primary headache" or "secondary headache"

SECONDARY OUTCOMES:
Mortality (yes/no) | Month 1
  "Mortality" refers to whether or not the subject is still alive.
Length of stay in the emergency department (days) | Month 1
Length of stay in the hospital (days) | Month 1
White blood cell count in cerebral spinal fluid | Month 1
Red blood cell count in cerebral spinal fluid | Month 1
Cerebral spinal fluid glucose level | Month 1
Cerebral spinal fluid protein level | Month 1
Cerebral spinal fluid chloride level | Month 1
Presence/absence of enterovirus in cerebral spinal fluid | Month 1
  Based on qualitative result from ELISA laboratory exam.
Presence/absence of herpes virus in cerebral spinal fluid | Month 1
  Based on qualitative result from ELISA laboratory exam.
Presence/absence of cerebral imaging indicating an ischemic or hemorrhagic stroke, subarachnoid hemorrhage, an expansive process, cerebral trombophlebitis cerebral or other abnormalities suggestive of a secondary cause of headache. | Month 1
Secondary headache onset: yes/no | Month 1
  Was there secondary headache onset by month 1?

CONTACTS AND LOCATIONS:
Overall Officials: Romain Genre Grandpierre, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Grau-Mercier L, Grandpierre RG, Alonso S, Savey A, Le Floch A, de Oliveira F, Masia T, Jory N, Coisy F, Claret PG. S100B serum level: A relevant biomarker for the management of non-traumatic headaches in emergency care? Am J Emerg Med. 2023 Jun;68:132-137. doi: 10.1016/j.ajem.2023.03.036. Epub 2023 Mar 25. PMID 37001377